CLINICAL TRIAL: NCT02335476
Title: Automatic Early Melanoma Detection by Ultrahigh Resolution Three Dimensional Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201402036RINA
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Melanoma
Keywords: optical coherence tomography
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will use optical coherence tomography to detect the ex-vivo tissue image of surgical removed melanoma or other benign pigmented lesions of skin.

DETAILED DESCRIPTION:
The investigators will use an advanced high resolution 3D optical coherence tomography (OCT) technology to observe skin tissue images in ex vivo culture. Parts of melanoma or benign pigmented lesions specimens derived from biopsy or surgical excision specimen will be observed by 3D optical tomography. A tiny tissue fragment of melanoma or benign pigmented lesions will be taken from surgical specimen without interference normal pathological evaluation. The location of melanocytic cells in melanoma or benign tissue fragments will be mapped by the 3D optical coherence tomography (OCT). The 3D optic tomography system utilize a Ce:YAG optical fiber as light source and also combined with confocal microscopy. Taken together, these features made the 3D optic tomography system have very high resolution and suitable for single cell imaging. This study will not interfere with the normal medical practice and had no impact on patient's safety and health. All of the materials will be destroyed once the experiments are done. The enrollment criteria will be dermatological patients who need to surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged older than 20 years old
* Patients who had melanoma, melanoma in situ, and/or other benign pigmented lesions,
* Patients who had non-melanoma skin cancers (basal cell carcinoma, or squamous cell carcinoma).
* Patients who had precancerous skin lesions (Bowen's disease, actinicc keratosis)

Exclusion Criteria:

• Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients at out-patient clinics or ward of Department of Dermatology, National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Ex vivo Tissue image. | 1 day
  Partial fragments of tissue specimens from melanoma, melanoma in situ, or other benign pigmented lesions will be used for imaging purpose by a optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: JENGWEI TJIU, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan